CLINICAL TRIAL: NCT04103203
Title: Fast Assay for Pathogen Identification - Quasi-Experimental Intervention Study
Acronym: FAPIC-QE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); School of Medicine, University of Zagreb (Unknown); Molzym (Unknown); AIT Austrian Institute of Technology GmbH (Other); BEE Robotics (Unknown); University of Warwick (Other); Claude Bernard University (Other); Axo Science (Unknown)
Responsible Party: Principal Investigator, prof. dr. Inge Gyssens, Prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19.51/Infect.19.02
Record Dates: First submitted 2019-07-12; First posted 2019-09-25 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Sepsis; Septic Shock; Bacteremia
MeSH Terms: conditions — Sepsis; Shock, Septic; Bacteremia

STUDY DESIGN:
Intervention Model Description: Quasi-experimental intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New diagnostic results NOT available (No Intervention): Patients with suspected sepsis are included. Blood samples will be collected and analysed with the new diagnostics. However, results will not be communicated. Only the results of routine blood cultures will be availabtle to the treating physician. No intervention will take place, care is provided according to normal routine practices.
- New diagnostic results available (Experimental): Patients with suspected sepsis are included. Blood samples will be collected and analysed with the new diagnostics. Results will be communicated via telephone by the consultant microbiologist and the electronic medical file to the treating physician. Results of routine blood cultures will also be available for all patients. Results of the new diagnostics are expected earlier, and the treating physician is able to make an earlier decision in terms of antibiotic therapy if he/she deems it necessary.
  Interventions: Diagnostic Test: PathoRobot/ Patho-Doc Test result

INTERVENTIONS:
Diagnostic Test: PathoRobot/ Patho-Doc Test result — Test results of the new diagnostics will be available to the treating physician.
  Arms: New diagnostic results available

SUMMARY:
The performance and clinical impact of two diagnostic systems will be evaluated using whole blood samples that are collected in parallel with samples for blood culture. As the rapid diagnostic systems will have the largest impact on severely ill patients (in need of a fast diagnosis) with bacterial infection, the evaluation will be performed in patients suspected of bacteraemia. During the study the new systems will be used in parallel with routine blood cultures. In alternating periods of 1 month, the results of the diagnostic system will be communicated to treating physicians (intervention) or not revealed (control). Blood culture results will be reported throughout the complete study period. Patients with suspected sepsis at the Emergency Department (ED), the department of infectious diseases/nephrology, and the department of haemodialysis will be included. In routine care, two blood culture sets (2x2 bottles) per patient are collected. One extra blood sample (EDTA tube, 9 ml of blood) will be sampled for each routine set of blood cultures. In addition, the clinical data of the patients will be collected. The samples will be sent to the clinical laboratory where samples are tested with the new systems during regular working hours in batches of 8 samples per run (2-3 runs per day). On average, 10%-20% of the blood cultures drawn on the presumption of bacteraemia yield bacterial pathogens. Previous data show that 13% of patients yield positive blood cultures. Thus, in order to collect blood samples of 100 new episodes of bacteraemia approximately 1000 patients (2000 blood cultures + 1000 EDTA tubes) have to be collected for each system (2000 patients in total). The results of the systems will be used to evaluate the clinical utility of the system regarding time to antibiotic treatment change and bacteraemia management. The system will be used directly for the diagnosis of patients, resulting in a possible change of treatment strategy. However, routine blood culture practices will still be done during the whole study period.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of sepsis
* The drawning of blood cultures
* Age >18 years

Exclusion Criteria:

* Children (<18 years)
* Patients who are not hospitalized and sent home after ED admission
* Duplicate blood cultures from the same bacteraemia episode (7days between positives with the same organism, or 24h for different organisms)
* Patients from who blood cultures are drawn on Friday evening (17h) or Saturday during intervention periods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1978 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Median time from specimen collection/arrival in the laboratory until antibiotic regimen change | at study completion, 10 months
  Time period between collection of blood cultures until the first change in antibiotic regimen

SECONDARY OUTCOMES:
Median time to appropriate, species-specific antibiotic therapy | at study completion, 10 months
  Time period between collection of blood cultures until the first administration of species-specific antibiotic therapy
In-hospital mortality | at study completion, 10 months
  In-hospital mortality
Time to organism identification | at study completion, 10 months
  Time period between collection of blood cultures until the time to identification of a causative organism with the new diagnostics and with blood cultures
Time to effective therapy | at study completion, 10 months
  Time period between collection of blood cultures until the first administration of antibiotic therapy effective againts the causative organism
Time to optimal therapy | at study completion, 10 months
  Time period between collection of blood cultures until the first administration of antibiotic therapy that is optimal for patient recovery
30-day all cause mortality | at study completion, 10 months
  Number of patients with 30-day all cause mortality
Length-of-stay | at study completion, 10 months
  Length of hospital stay
Length of ICU stay | at study completion, 10 months
  Length of stay in an Intensive Care Unit
Destination at Discharge | at study completion, 10 months
  Destination after discharge (home, rehabilitation home, nursing home, ...)

CONTACTS AND LOCATIONS:
Overall Officials: Inge C Gyssens, MD, PhD, Principal Investigator — Hasselt University
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605